CLINICAL TRIAL: NCT06490523
Title: Analysis of Advanced Physiological Ventilatory Parameters During Spontaneous Breathing Effort in Patients with Acute Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Principal Investigator, Andrea Castellvi, Clinical Investigator, Hospital del Mar
Other Study IDs: 2021/9742
Record Dates: First submitted 2024-06-25; First posted 2024-07-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Hypoxic Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICU survivors: Acute hypoxemic respiratory failure patients on invasive mechanical ventilation who survive to ICU discharge
- ICU non-survivors: Acute hypoxemic respiratory failure patients on invasive mechanical ventilation who do not survive to ICU discharge

SUMMARY:
The aim of this prospective physiological cohort study conducted in a medical intensive care unit (ICU) at Hospital del Mar in Barcelona, Spain, was to analyze the proportion of time spent within the "safe" range of respiratory effort (including esophageal pressure swing (ΔPes), respiratory muscular pressure (Pmus), and transdiaphragmatic pressure swing (ΔPdi)) in patients with acute hypoxemic respiratory failure (AHRF) undergoing invasive mechanical ventilation (IMV), during the active breathing phase in relation to ICU survival.

The investigators hypothesized that AHRF patients on IMV with better outcome (i.e., ICU survivors) spend more time within the "safe" range of respiratory effort during the active breathing phase compared to non-survivors.

AHRF patients on IMV were continuously monitored with esophageal and gastric manometry from the detection of the onset of respiratory effort for up to 7 days, or until extubation, or until death, whichever occurred first.

DETAILED DESCRIPTION:
To characterize in detail the evolution of respiratory effort over time, the investigators conducted a prospective observational cohort study with continuous recordings of airway pressure, flow, esophageal and gastric pressures for up to 7 days after the onset of respiratory effort in AHRF patients on IMV.

Patients were classified into two groups: ICU survivors and ICU non-survivors. The primary objective of the study was to analyze the proportion of time spent within a specified "safe" range for Pmus, ΔPes, and ΔPdi (respiratory effort physiological variables), during spontaneous breathing, comparing both groups during the first 7 days after the initiation of respiratory effort. The secondary objective was to analyze the median values of ΔPes, Pmus, and ΔPdi during the monitorization period (active breathing phase) between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypoxemic respiratory failure patients requiring invasive mechanical ventialtion

Exclusion Criteria:

* Presence of chest drains
* Contraindication to esophageal catheterization (e.g., recent upper gastrointestinal surgery, bleeding esophageal varices)
* Concomitant acute exacerbation of obstructive airways disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older who were admitted to the ICU and required invasive mechanical ventilation (IMV) for acute hypoxemic respiratory failure (AHRF) were eligible for the study. Patients were excluded if they had chest drains, a contraindication to esophageal catheterization (e.g., recent upper gastrointestinal surgery, bleeding esophageal varices), or a concomitant acute exacerbation of obstructive airways disease.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of time spent in different ranges of ΔPes (low, safe, and high) during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  The defined "safe" range for ΔPes was -5 to -10 cm H2O. Effort outside the defined "safe" range was categorized as "low" if it fell below the lower limit, or "high" if it exceeded the upper limit of the safe range for the variable.
Proportion of time spent in different ranges of Pmus (low, safe, and high) during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  The defined "safe" range for Pmus was 5 to 15 cm H2O. Effort outside the defined "safe" range was categorized as "low" if it fell below the lower limit, or "high" if it exceeded the upper limit of the safe range for the variable.
Proportion of time spent in different ranges of ΔPdi (low, safe, and high) during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  The defined "safe" range for ΔPdi was 3 to 12 cm H2O. Effort outside the defined "safe" range was categorized as "low" if it fell below the lower limit, or "high" if it exceeded the upper limit of the safe range for the variable.
Median value of ΔPes during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  To analyze the median value of ΔPes during the active breathing phase between the two groups in cm H20.
Median value of Pmus during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  To analyze the median value of Pmus during the active breathing phase between the two groups in cm H20.
Median value of ΔPdi during the active breathing phase between the two groups | From the start the start of respiratory effort up to 7 days (or until extubation or death, if earlier)
  To analyze the median value of ΔPdi during the active breathing phase between the two groups in cm H20.

SECONDARY OUTCOMES:
The need for the use of venovenous (VV) extracorporeal membrane oxygenation (ECMO) | From date of initiation of invasive mechanical ventilation until extubation or date of death from any cause, whichever came first, assessed up to 24 months
  Initiation of VV ECMO during the mechanical ventilation period (yes or no)
The need for the use of extracorporeal CO2 removal (ECCO2R) | From date of initiation of invasive mechanical ventilation until extubation or date of death from any cause, whichever came first, assessed up to 24 months
  Initiation of ECCO2R during the mechanical ventilation period (yes or no)
The need for a Tracheostomy | From date of initiation of invasive mechanical ventilation until extubation or date of death from any cause, whichever came first, assessed up to 24 months
  The need to perfom a tracheostomy duduring the mechanical ventilation period (yes or no)
Duration of invasive mechanical ventilation (IMV) | From date of initiation of invasive mechanical ventilation until extubation or date of death from any cause, whichever came first, assessed up to 24 months
  Duration of IMV measured in days
Intensive care Unit (ICU) Length of stay | From date of ICU admission until date of ICU discharge or date of death from any cause, whichever came first, assessed up to 24 months
  Duration of the ICU admission measured in days
Hospital Length of stay | From date of Hospital admission until date of Hospital discharge or date of death from any cause, whichever came first, assessed up to 24 months
  Duration of the Hospital admission measured in days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Telias I, Brochard LJ, Gattarello S, Wunsch H, Junhasavasdikul D, Bosma KJ, Camporota L, Brodie D, Marini JJ, Slutsky AS, Gattinoni L. The physiological underpinnings of life-saving respiratory support. Intensive Care Med. 2022 Oct;48(10):1274-1286. doi: 10.1007/s00134-022-06749-3. Epub 2022 Jun 12. PMID 35690953
- [Background] Sklar MC, Madotto F, Jonkman A, Rauseo M, Soliman I, Damiani LF, Telias I, Dubo S, Chen L, Rittayamai N, Chen GQ, Goligher EC, Dres M, Coudroy R, Pham T, Artigas RM, Friedrich JO, Sinderby C, Heunks L, Brochard L. Duration of diaphragmatic inactivity after endotracheal intubation of critically ill patients. Crit Care. 2021 Jan 11;25(1):26. doi: 10.1186/s13054-020-03435-y. PMID 33430930
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. Spontaneous breathing during lung-protective ventilation in an experimental acute lung injury model: high transpulmonary pressure associated with strong spontaneous breathing effort may worsen lung injury. Crit Care Med. 2012 May;40(5):1578-85. doi: 10.1097/CCM.0b013e3182451c40. PMID 22430241
- [Background] Goligher EC. Myotrauma in mechanically ventilated patients. Intensive Care Med. 2019 Jun;45(6):881-884. doi: 10.1007/s00134-019-05557-6. Epub 2019 Feb 11. No abstract available. PMID 30741329
- [Background] Goligher EC, Brochard LJ, Reid WD, Fan E, Saarela O, Slutsky AS, Kavanagh BP, Rubenfeld GD, Ferguson ND. Diaphragmatic myotrauma: a mediator of prolonged ventilation and poor patient outcomes in acute respiratory failure. Lancet Respir Med. 2019 Jan;7(1):90-98. doi: 10.1016/S2213-2600(18)30366-7. Epub 2018 Nov 16. PMID 30455078
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Kondili E, Alexopoulou C, Xirouchaki N, Vaporidi K, Georgopoulos D. Estimation of inspiratory muscle pressure in critically ill patients. Intensive Care Med. 2010 Apr;36(4):648-55. doi: 10.1007/s00134-010-1753-4. Epub 2010 Jan 28. PMID 20107765
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Jonkman AH, Telias I, Spinelli E, Akoumianaki E, Piquilloud L. The oesophageal balloon for respiratory monitoring in ventilated patients: updated clinical review and practical aspects. Eur Respir Rev. 2023 May 17;32(168):220186. doi: 10.1183/16000617.0186-2022. Print 2023 Jun 30. PMID 37197768
- [Background] Chiumello D, Consonni D, Coppola S, Froio S, Crimella F, Colombo A. The occlusion tests and end-expiratory esophageal pressure: measurements and comparison in controlled and assisted ventilation. Ann Intensive Care. 2016 Dec;6(1):13. doi: 10.1186/s13613-016-0112-1. Epub 2016 Feb 12. PMID 26868503
- [Background] Goligher EC, Dres M, Patel BK, Sahetya SK, Beitler JR, Telias I, Yoshida T, Vaporidi K, Grieco DL, Schepens T, Grasselli G, Spadaro S, Dianti J, Amato M, Bellani G, Demoule A, Fan E, Ferguson ND, Georgopoulos D, Guerin C, Khemani RG, Laghi F, Mercat A, Mojoli F, Ottenheijm CAC, Jaber S, Heunks L, Mancebo J, Mauri T, Pesenti A, Brochard L. Lung- and Diaphragm-Protective Ventilation. Am J Respir Crit Care Med. 2020 Oct 1;202(7):950-961. doi: 10.1164/rccm.202003-0655CP. PMID 32516052
- [Background] Carteaux G, Mancebo J, Mercat A, Dellamonica J, Richard JC, Aguirre-Bermeo H, Kouatchet A, Beduneau G, Thille AW, Brochard L. Bedside adjustment of proportional assist ventilation to target a predefined range of respiratory effort. Crit Care Med. 2013 Sep;41(9):2125-32. doi: 10.1097/CCM.0b013e31828a42e5. PMID 23787397
- [Background] de Vries H, Jonkman A, Shi ZH, Spoelstra-de Man A, Heunks L. Assessing breathing effort in mechanical ventilation: physiology and clinical implications. Ann Transl Med. 2018 Oct;6(19):387. doi: 10.21037/atm.2018.05.53. PMID 30460261
- [Derived] Parrilla-Gomez FJ, Castellvi-Font A, Boutonnet V, Parrilla-Gomez A, Antolin Terreros M, Mestre Somoza C, Blanes Bravo M, Pratsobrerroca de la Rubia P, Martin-Lopez E, Marco S, Festa O, Brochard LJ, Goligher EC, Masclans Enviz JR. Association of Breathing Effort With Survival in Patients With Acute Respiratory Distress Syndrome. Crit Care Med. 2025 Oct 1;53(10):e1982-e1994. doi: 10.1097/CCM.0000000000006797. Epub 2025 Aug 5. PMID 40758388